CLINICAL TRIAL: NCT04445246
Title: Inhaled Iloprost for the Treatment of Suspected COVID-19 Respiratory Failure
Brief Title: Inhaled Iloprost for Suspected COVID-19 Respiratory Failure
Acronym: ILOCOVID
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hamad Medical Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MRC-05-026
Record Dates: First submitted 2020-06-09; First posted 2020-06-24 (Actual); Last update posted 2022-03-29 (Actual); Status verified 2020-05

CONDITIONS: COVID-19; ARDS, Human; Hypoxemic Respiratory Failure
Keywords: Iloprost; prostacyclins; inhaled nitric oxide; pulmonary vasodilators
MeSH Terms: conditions — COVID-19; Respiratory Distress Syndrome; Respiratory Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Inhaled Iloprost therapy (Experimental): Inhaled Iloprost 20 mcg every 8 hours for 5 days only delivered by nebulization
  Interventions: Drug: Inhaled ILOPROST

INTERVENTIONS:
Drug: Inhaled ILOPROST — Inhaled Iloprost 20 mcg every 8 hours for 5 days only delivered by nebulization.
  Other Names: Ventavis by Actelion Pharmaceuticals US, Inc.

SUMMARY:
Acute respiratory distress syndrome (ARDS) is a type of respiratory failure characterized by the rapid onset of widespread inflammation in the lungs. ARDS is thought to be the main cause of respiratory failure in COVID-19 patients. Research is still ongoing to further elucidate the different ARDS subtypes that may exist in COVID-19. It is crucial to find new targets for treatment and support of COVID-19 patients with respiratory failure.

DETAILED DESCRIPTION:
The investigators hypothesize that inhaled prostacyclins (Iloprost in this study) may improve inflammation and oxygenation in suspected or confirmed COVID-19 patients with respiratory failure.

Research participants: Suspected or confirmed COVID-19 patients presenting to the emergency department (ED) of intensive care units (ICU) with Hypoxemic respiratory failure.

Intervention: Inhaled Iloprost (Tradename Ventavis by Actelion Pharmaceuticals US, Inc.) three times daily for 5 days Methods: patients will be screened in ED and ICU for inclusion and exclusion criteria and then consent will be obtained. The intervention will be started within 48 hours of presentation. Baseline parameters on oxygenation, inflammatory markers, hemodynamics will be obtained and followed serially over the period of the intervention. Additional data about time to intubation, time on mechanical ventilation, lung mechanics, and need for prone positioning will also be collected.

Data will be analyzed for percentage improvement in oxygenation (Oxygen saturation and PaO2/FiO2 ratio), trends of inflammatory markers, and hemodynamic stability while Iloprost is administered.

Based on previous studies of Iloprost on ARDS patients, the investigators anticipate an improvement in oxygenation and inflammatory parameters and possible prevention of intubation with shorter mechanical ventilation times. Iloprost showed a safe profile with stable hemodynamics during administration.

ELIGIBILITY:
Inclusion Criteria:

1. Suspected or confirmed COVID-19 patient by PCR
2. O2 saturation =<92% on 5 or more l/min of O2 by NC or Face mask
3. On CPAP, HFNC or Invasive ventilation
4. Enrollment within 48h of onset of hypoxemia

Exclusion Criteria:

1. Age <18
2. Pregnancy or Positive pregnancy test at the time of screening
3. Clinical evidence of left atrial hypertension or known chronic CHF
4. Persistent Hypotension SBP<85 on presentation
5. Mechanical ventilation >7 days
6. Patients who received iloprost treatment for any indication within 48 hours prior to enrollment in the clinical trial or patients who were on thrombin inhibitors, or nitric oxide within the previous 24 h before study randomization are also excluded.
7. Patients with contraindication for ilioprost

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2020-05-23 (Actual); Primary Completion 2021-05-31 (Actual); Study Completion 2021-05-31 (Actual)

PRIMARY OUTCOMES:
change in oxygenation parameters | 5 days
  change in oxygen saturation and PaO2/FiO2 ratio by 20% on day 6 compared to baseline values prior to Iloprost initiation.

SECONDARY OUTCOMES:
Rates of endotracheal intubation | 28 days
  likelihood to require intubation in the cohort treated with Iloprost
Invasive ventilation duration | 28 days
  in days in the cohort treated with Iloprost
ICU length of stay | 28 days
  in days in the cohort treated with Iloprost
Hospital Length of stay | 28 days
  in days in the cohort treated with Iloprost
Rates of proning therapy | 28 days
  likelihood to require proning in the cohort treated with Iloprost
Rates of ECMO cannulation | 28 days
  likelihood to require ECMO cannulation in the cohort treated with Iloprost
Mortality | 28 days
  likelihood to die of any cause within 28 days of initial hospital presentation

CONTACTS AND LOCATIONS:
Overall Officials: Nadir Kharma, MD, Principal Investigator — Hamad Medical Corporation
Locations (1):
- Hamad Medical Corporation, Doha, Qatar

REFERENCES:
- [Derived] Mulia EPB, Luke K. Inhaled prostacyclin analogues in COVID-19 associated acute respiratory distress syndrome: scientific rationale. Egypt Heart J. 2021 Sep 16;73(1):82. doi: 10.1186/s43044-021-00208-y. PMID 34529182